CLINICAL TRIAL: NCT06784024
Title: Topical Lidocaine vs. Traditional Management in Manual Vacuum Aspiration Pain Management, for Endometrial Thickness. Randomized Double-blind Clinical Trial.
Brief Title: Topical Lidocaine vs. Traditional Management in Manual Vacuum Aspiration Pain Management.
Acronym: ENDOLID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ricardo A Gutierrez Ramirez, MD, MSc, FACOG (Other)
Responsible Party: Sponsor-Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Titular professor, Universidad Nacional Autonoma de Honduras
Organization: Universidad Nacional Autonoma de Honduras (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGO-UNAH-48-1-2025
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-02

CONDITIONS: Endometrial Hyperplasia; Endometrial Diseases
Keywords: Lidocaine; manual vacuum aspiration; Pain management
MeSH Terms: conditions — Endometrial Hyperplasia; Uterine Diseases; Agnosia | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel-group (Group A and Group B) clinical trial of superiority and efficacy.
Who Masked: Participant, Investigator
Masking Description: Randomization ensures that participants are equally distributed between treatment groups (topical lidocaine and placebo), which minimizes selection bias and confounding. This allows observed differences in outcomes to be attributed to treatment rather than other variables.
  - Double Blind: Keeping both participants and investigators uninformed regarding the treatment group eliminates observer bias and patient expectation bias. This is crucial for obtaining valid and objective results on the effectiveness of topical lidocaine in pain management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Experimental): Topical lidocaine (SPRAY SOLUTION 10 g) 10% will be applied to the cervix and cervical canal prior to the MVA procedure in a number of 20 sprays separated by 3 seconds between each spray (0.06 ml/spray).
  Interventions: Drug: Lidocaine topical
- Control (Placebo Comparator): Placebo (0.9% saline) will be applied topically to the cervix and cervical canal prior to the MVA procedure in a number of 20 sprays separated by 3 seconds between each spray (0.06 ml / spray).
  Interventions: Other: Saline solution

INTERVENTIONS:
Drug: Lidocaine topical — Topical lidocaine (SPRAY SOLUTION 10 g) 10% will be applied to the cervix and cervical canal prior to the MVA procedure in a number of 20 sprays separated by 3 seconds between each spray (0.06 ml/spray).
  Other Names: Lidocaine
  Arms: Lidocaine
Other: Saline solution — Placebo (0.9% saline) will be applied topically to the cervix and cervical canal prior to the MVA procedure in a number of 20 sprays separated by 3 seconds between each spray (0.06 ml / spray).
  Other Names: SSN 0.9%
  Arms: Control

SUMMARY:
The main objective of this study is to evaluate the effect of lidocaine versus placebo according to the visual analog pain scale, during manual uterine aspiration in patients with endometrial thickening, by means of a prospective, randomized, double-blind, placebo-controlled clinical trial, taking into account women with a diagnosis of endometrial thickening, requiring MVA, which will be performed in the emergency area of Obstetrics and Gynecology of the Hospital Materno Infantil, by resident physicians of the second year of the residency of said postgraduate course supervised by specialist physicians. A sample of 126 participants will be studied, divided into 2 groups of 63 patients each (control and intervention), the first group will be given placebo and the second group will be given lidocaine 10%, 20 sprays, in addition to the pre-established pain management for MVA, and the pain perception before, during and after the procedure will be evaluated by means of the visual analog pain scale. The data will be tabulated and analyzed in Redcap (software) using descriptive statistics.

DETAILED DESCRIPTION:
The Manual Vacuum Aspiration (MVA) procedure consists of extracting residual or retained tissues from the uterine cavity through a cannula connected to a portable aspirator that creates a manual vacuum. It is characterized for being simple, safe, effective and accepted by patients, since it is economical, fast and does not require hospitalization in comparison to "Instrumental Uterine Curettage".

Worldwide, abnormal uterine bleeding, endometrial thickening and abortion are considered a public health problem. These conditions put women's lives at risk and because of this, the manual vacuum aspiration technique (MVA) was developed to provide more humane care to women who come to hospitals for incomplete abortions. MVA uses flexible plastic hoses (Karman) of various sizes (4 to 12 mm). It can be adapted to the woman's needs, eliminating the need to dilate the cervix.

Among the important points to consider for the performance of this protocol is pain management, which, in a standardized way, is treated with paracervical block with local anesthesia, which is an effective method for pain management and should be part of all vacuum aspiration procedures. This, considering that about 97% of women who undergo it report pain during and after the procedure. Therefore, non-steroidal anti-inflammatory drugs are also widely used 30 minutes prior to the procedure.

In a Swedish study of 200 patients who underwent MVA for incomplete abortion and uterine size less than eight weeks gestation, patients were allowed to choose between general anesthesia or paracervical block. Of the 37 patients who chose MVA with paracervical block, none requested conversion to general anesthesia. Therefore, it can be deduced that there are satisfactory results with paracervical block.

Studies in Latin America have shown that Manual Vacuum Aspiration is a safe technique, clinically effective, fast, with less blood loss and less painful than LUI. Mexico and Colombia are two of the countries that use this technique the most, since it has been shown to be less associated with complications, such as uterine perforation, hemorrhage, infections and traumatic injuries that may exist in comparison with instrumental curettage. In several studies, the effectiveness of MVA has been shown to be greater than 98%.

It should be noted that MVA has proven to be a highly effective and safe procedure, even at the first level of care. Most women recover within a few hours.

In Honduras, the Women's Rights Center describes MVA as a considerable alternative to curettage, because it is safer and just as effective, without the need for general anesthesia, and can be performed in healthcare settings that are not strictly hospitals, for example, in health centers, if trained professionals are available. This allows the optimization of limited resources and a significant increase in women's access to treatment services. It is worth mentioning that the recovery period is shorter, so there is a substantial saving in the occupation of beds and hospital supplies and the time of incapacity is reduced in each patient.

MVA is considered by both the WHO and FIGO to be modern, versatile, safe and effective as long as the personnel trained in this medical technique and the correct equipment are available.

Pain management is an important aspect to consider when carrying out this procedure, which is why this study has special relevance, since, in our country, it constitutes one of the main treatment options for several gynecological-obstetric conditions, as it is a cost-effective tool that optimizes available resources. To know if there is any change when using topical lidocaine vs. placebo in a double-blind study, this, as a coadjuvant to standardized management, would significantly broaden the perspective and the knowledge we have about this practice, giving the possibility of improving the quality of the service offered by the hospital centers, by knowing the reality regarding the patient's perception of pain and being able to offer new analgesia alternatives or also, it is possible to contemplate the possibility of reducing costs in the performance of the procedure. Therefore, we consider that it would be very useful to obtain the results of this research, in addition to the fact that there are no related studies in the region.

ELIGIBILITY:
Inclusion Criteria:

* Be in good general health, as evidenced by your medical history, or have been diagnosed with endometrial thickening or have abnormal uterine bleeding.
* Ultrasonography with endometrial line greater than 5 mm
* Normotensive
* Over 40 years of age
* Able to give informed consent to participate in the study.
* Cervical dilatation > 2 mm
* Cervical dilatation < 10 mm
* Patient without hemodynamic decompensation.
* Submission of a signed and dated informed consent form.
* Declared willingness to comply with all study procedures and availability for the duration of the study.
* Menopausal woman.
* Willingness to comply with the protocol regimen.
* Possess a cell phone.
* Ability to read.
* Know how to write.
* To reside in Francisco Morazán.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patients with severe cardiovascular diseases.
* Presence of active gynecological infections.
* History of severe adverse reactions to lidocaine.
* Acute pelvic pain.
* Mental disability preventing informed consent.
* Hemodynamic decompensation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | Since intervention until 2 hours
  It is a horizontal line of 10 centimeters, at the ends of which the extreme expressions of a symptom are shown. On the left side is located the absence or lower intensity and on the right side the higher intensity. The patient is then asked to mark on the line the point indicating the intensity and it is measured with a millimeter ruler. The intensity is expressed in centimeters or millimeters.
  The scale will be measured at 5 times:
  During the administration of injectable lidocaine During the placement of the Pozzi clamp During the introduction of the cannula 120 seconds after starting the procedure 2 hours after starting the procedure

SECONDARY OUTCOMES:
Adverse effects of lidocaine | Since intervention until 24 hours
  incidence of Adverse effects of lidocaine

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Gutierrez Ramirez, MD, MSc, Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No
It is not necessary, none of the 18 HIPAA identifiers will be placed

REFERENCES:
- [Background] Charoenkwan K, Nantasupha C. Methods of pain control during endometrial biopsy: A systematic review and meta-analysis of randomized controlled trials. J Obstet Gynaecol Res. 2020 Jan;46(1):9-30. doi: 10.1111/jog.14152. Epub 2019 Oct 30. PMID 31667985